CLINICAL TRIAL: NCT01259076
Title: Effect of Weight Loss on Breast Density Using Both Digital Mammography and Breast MRI
Brief Title: Effect of Weight Loss on Breast Density Using Digital Mammography and MRI in Women Who Are At Increased Risk For Breast Cancer
Status: Terminated | Type: Observational
Why Stopped: Study was closed early due to slow accrual.
Sponsor: Northwestern University (Other)
Collaborators: Robert H. Lurie Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: NU 10B01; STU00038177 (Other: Northwestern University IRB)
Record Dates: First submitted 2010-12-10; First posted 2010-12-13 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Healthy, no Evidence of Disease
MeSH Terms: interventions — Magnetic Resonance Spectroscopy; Surgical Procedures, Operative; Congresses as Topic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group 1: Participants who are eligible for and have opted to undergo gastric bypass surgery
  Interventions: Procedure: magnetic resonance imaging; Procedure: digital mammography; Procedure: conventional surgery
- Group 2: Participants who are eligible for but decided not to undergo gastric bypass surgery.
  Interventions: Procedure: magnetic resonance imaging; Procedure: digital mammography

INTERVENTIONS:
Procedure: magnetic resonance imaging — Undergo MRI at baseline and 1 year later.
  Other Names: MRI; NMR imaging; NMRI; nuclear magnetic resonance imaging
Procedure: digital mammography — Undergo digital mammography at baseline and 1 year later.
Procedure: conventional surgery — Undergo gastric bypass surgery
  Other Names: surgery, conventional
  Groups: Group 1

SUMMARY:
Diagnostic procedures, such as digital mammography and MRI, may help measure how weight loss affects breast density in women who are at increased risk for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. To determine if weight loss in patients undergoing Roux en Y gastric bypass procedures has any effect on breast density as measured by mammography and breast MRI. OUTLINE: GROUP I: Participants undergo mammography and MRI at baseline and 1 year. Participants also undergo gastric bypass surgery. GROUP II: Participants undergo mammography and MRI at baseline and 1 year. After completion of study treatment, patients are followed up at 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Women eligible for gastric bypass surgery
* Pre-menopausal women
* All women will have signed an informed consent form prior to participating in study procedures

Exclusion Criteria:

* Women with a history of breast cancer
* Women currently taking exogenous hormone replacement therapy
* Women currently taking a SERM
* Women currently taking an aromatase inhibitor
* Pregnant or lactating women
* Women who have been pregnant or lactating in the past 2 years
* Women who have metallic or other surgical implants
* All subjects will have a determination of their estimated glomerular filtration rate (eGFR) within 24 hours of undergoing any study where gadolinium based contrast agents will be administered
* Subjects should not have a known history of recent onset acute renal dysfunction
* Subjects with a history of stable chronic renal dysfunction may participate in studies using GBCA based on their eGFR, as outlined below
* Subjects should not have severe liver dysfunction, particularly when associated with kidney disease
* Subjects should receive GBCAs in the perioperative period (i.e. within 4 weeks) after renal or liver transplantation

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pre-menopausal women between the ages of 30 and 50 who are eligible and undergoing evaluation for gastric bypass surgery
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2011-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in BMI and breast density | At baseline and year 1

CONTACTS AND LOCATIONS:
Overall Officials: Nora Hansen, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States